CLINICAL TRIAL: NCT03194997
Title: Pilates and Dance to Breast Cancer Patients Undergoing Treatment: MoveMama Project
Brief Title: Pilates and Dance to Breast Cancer Patients Undergoing Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratório de Pesquisa em Lazer e Atividade Física (Other)
Collaborators: Centro de Pesquisas Oncológicas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2.073.549
Record Dates: First submitted 2017-06-16; First posted 2017-06-22 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer; Quality of Life; Lymphedema; Fatigue; Depressive Symptoms; Body Image; Self Esteem; Optimism; Sexual Function Disturbances; Stress; Sleep Disturbance; Pain; Muscular Weakness; Postural Balance; Range of Motion; Cardiorespiratory Fitness
Keywords: Breast Cancer; Quality of life; Lymphedema; Fatigue; Depressive symptoms; Body image; Self Esteem; Optimism; Sexual function; Stress; Sleep quality; Pain; Muscular strength; Postural; Balance; Range of motion; Cardiorespiratory fitness
MeSH Terms: conditions — Breast Neoplasms; Lymphedema; Fatigue; Depression; Sexual Dysfunctions, Psychological; Parasomnias; Pain; Muscle Weakness; Sleep Initiation and Maintenance Disorders | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial, three-arm study (group 1 - Dance; group 2 - Pilates and group 3 - Control), single-blinded.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dance (Experimental): The group randomized to Dance intervention will receive a 3-week intervention with belly dance classes. The classes will be divided in: Warm up and stretching (10 minutes), Main part with belly dance steps and movements (40 minutes) and relaxation (10 minutes).
  Interventions: Other: Dance
- Pilates (Experimental): The group randomized to Pilates intervention will receive a 3-week intervention with Pilates Methods. The classes will be divided in: Warm up and stretching (10 minutes), Main part with Pilates exercises (40 minutes) and relaxation (10 minutes).
  Interventions: Other: Pilates
- Control (No Intervention): The group randomized to Control group will be invited to maintain routine activities and be contacted by phone every two months and will receive an explanatory booklet on the benefits of physical activity after diagnosis of breast cancer as well as instructions on lymphedema prevention. Also, this group will be invited to three meeting during the 16 weeks of intervention, the first meeting will focus on stretching exercise to develop at home, a second meeting will be about self-esteem and the last meeting will be about prevented of lymphedema. The women in this group will not receive a dance or pilates intervention.

INTERVENTIONS:
Other: Dance — The Dance intervention will be performed with belly dance methods. It will occur 3 times per week, during 16 weeks, with 60 minutes the session.
  Arms: Dance
Other: Pilates — The Pilates intervention will be performed using specific exercises of Pilates Methods. During the classes it will be used thera band, toning ball and pilates ball. It will occur 3 times per week, during 16 weeks, with 60 minutes the session.
  Arms: Pilates

SUMMARY:
Breast cancer is one of the most common types of cancer in Brazil, and its treatment, namely surgery, chemotherapy, radiotherapy or hormone therapy, has consequences and side effects that significantly affect the quality of life and associated physical and psychological factors. The practice of physical activity, in turn, may play a beneficial role in these factors, and help the recovery of the patient in relation to the consequences of the treatments. Two types of physical activity can be addressed in the context of breast cancer; Dance and the Pilates method. Thus, the objective of the present study will be to analyze the impact of Pilates practice and dance on quality of life and on psychological and physical factors in patients undergoing adjuvant treatment of breast cancer. Patients older than 18 years who are in adjuvant treatment, namely, chemotherapy, radiotherapy and / or hormone therapy at the Oncology Research Center - CEPON, will be invited to be part of the study. With a randomized clinical trial of three arms, the patients will be submitted to 16 weeks of intervention, and randomized in 3 groups: (A) belly dance protocol group; (B) Pilates method protocol group, and (C) control group who will continue with their routine activities. Sample randomization will be conducted in confidence by one of the researchers in a specific computer program. Information about personal and clinical characteristics, quality of life, psychological factors (depressive symptoms, body image, self-esteem, optimism, perceived stress, fatigue, pain, sexual function and sleep quality) and physical factors (cardiorespiratory fitness, balance , Posture, upper limb functionality and presence of lymphedema). All information will be collected before and after the intervention period. Statistical analysis will use the statistical package SPSS - IBM, version 20.0. Firstly, descriptive statistics (mean, standard deviation and percentage) will be used in order to know the data, and then the Anova two way test with repeated measurements and Sydak Comparison Test, in order to analyze the data. Groups of the Pilates method, of the dance and control group. Significance level of 5%.

DETAILED DESCRIPTION:
The MoveMama Project includes two protocols: (1) Dance and (2) Pilates. Each session for each modality will last 60 minutes, three times a week, for 16 weeks.

In both groups, a chart of patient evolution will be developed during the protocol, which should be updated every week by the researchers responsible for the intervention. In order to control the intensity and safety of the practice of physical activity, since they are about patients who are in period of clinical adjuvant treatment. In this way, the blood pressure (BP), through a sphygmomanometer, and the investigation of the heart rate (HR) will be performed in every first class of the week at the beginning and end of the session.

The Subjective Effort Perception Scale - Borg Scale 6-20 points (BORG, 2000) will also be used to evaluate the intensity and / or discomfort during physical activity practice in both protocols. This 6 to 20-point scale can be used efficiently because of its relationship to heart rate. It should be applied to describe resting sensations to situations of maximum physical effort, considering number six equivalent to 60 bpm (beats per minute), as well as number 20 to 200 bpm (Table 2) (FOSS et al., 2000).

In both modalities of intervention, the evolution of the movements of upper limbs will always be respecting the limit of each patient.

The dance protocol (1) will be performed through the belly dance method. This type of methodology was selected, because it is a practice that involves an intimate relationship between movement and emotion, awakens a spontaneous body language that privileges movements that respect the individuality of each practitioner, for the recovery of the feminine identity, and for be a practice that proposes intense movements of the upper limbs, benefiting patients directly.

Classes will proceed in the following order: (a) Initial stretching: The sequence of movements lesson will span wide to specific joint movements, including flexion, extension, abduction, adduction and rotation, initiated by the upper body until reaching the lower limbs, with an expected duration of 10 minutes. (b) Main part: brief explanations about the purpose of the lesson, that is, the theory of dance or the specific step to be worked, followed by the practical part of teaching the technique. The purpose of this moment will be to develop in the students the movements of the belly dance technique, stimulating the motor coordination, the rhythm and the corporal consciousness, improving aspects of the flexibility and the range of movement of the upper limb. The practice of the movements will be explored in individual dynamics, in double or in group, involving the movement according to the rhythm of the music, or also, by rhythms stipulated by the students. This class session will last an average of 40 minutes. (c) Relaxation: Developed from slow-moving practices. With normalization of cardiac frequency, this part will last 10 minutes. Finally, at the end of each class, a brief discussion will be carried out on each student's perception of the contents given, and in relation to the objectives discussed at the beginning of the lesson, whether they were reached or not.

The Pilates protocol (2) will proceed in the following order: (a) Initial stretching: The breathig, imprint & release, hip release, spinal rotation, cat stretch, hip rolls, scapula isolation, arm circles, head nods and elevation & depression of scapulae exercises will be performed during warm-up in all sessions, then in the 10th session Added theraband, tonning ball and ball, intensifying the exercises. Duration of 10 minutes. (b) Main part: brief explanations about the purpose of the lesson, the theory of Pilates, the basic principles of Joseph Pilates: breathing, centering, control, precision, fluency and concentration. Clarify the positions: positioning of the pelvis, positioning of the rib cage, stabilization and movement of the shoulder girdle and positioning of the head and cervical spine. This part will include the specific exercises in Pilates. The practice of the movements will be explored in individual dynamics. This class session will last an average of 40 minutes. (c) Relaxation: The relaxation will consist of the exercises: sitting on the ball, sitting on the spine stretch forward ball, sitting on the self-stretching ball of the cervical muscles (Upper Trapezius and Muscle Scalene muscles) and active mobilization of the cervical spine during the 48 sessions. Duration of 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Stage I to III of breast cancer;
* Be in adjuvant treatment with chemotherapy, radiation therapy or hormone therapy;
* Receive the release of the oncologist responsible for the practice of physical activity, as well as the Physical Therapy Sector of CEPON.

Exclusion Criteria:

* Present some orthopedic or neurological limitation that not allows the practice of physical activity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Perception of Quality of life | 10 minutes
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30 and BR23). Scores range from zero to 100, and the higher the score, the better the quality of life on functional and general health scales, and the smaller the score, worse is the quality of life on the symptomatic scale.

SECONDARY OUTCOMES:
Depressive Symptoms | 10 minutes
  Beck's Depression Inventory - The scores goes from 0 to 63, and the higher score indicates more presence of depressive symptoms.
Body image | 10 minutes
  Body Image After Breast Cancer (BIBCQ) - Scores 0 to 45. Higher the score worst is the body image.
Self-Esteem | 5 minutes
  Rosenberg Self Esteem Scale - Scores 0 to 40 points. Higher the score better is the self-esteem.
Optimism | 5 minutes
  Life Orientation Test - (LOT-R) 0 to 40. It is determined that the higher the score, the greater the patients' optimism.
Stress | 5 minutes
  Perceived Stress Scale - Scores 0 to 56 points. Higher scores are associated with greater perceived stress.
Fatigue | 5 minutes
  Functional Assessment of Cancer Therapy-Fatigue (FACT-F) - Scores 0 to 52, a higher score indicates a level of less perceived fatigue.
Sexual function | 10 minutes
  Female Sexual Function Index (FSFI) - Scores 2 to 36 points, considering that the higher the score obtained, the better the sexual function of the woman.
Sleep Quality | 10 minutes
  Pittsburgh Sleep Quality Index - Scores 0 to 21, scores up to five determine a quality sleep ball, and scores greater than five points distinguish poor sleep quality.
Pain level | 3 minutes
  Visual Analog Scale - 0 to 10 points. Nearer to 10 indicates more pain.
Cardiorespiratory fitness | 10 minutes
  Six-Minute Walk Test - Vo2max estimation
Physical Activity | 10 minutes
  International Physical Activity Questionnaire - sedentary; insufficiently active; and very active and minutes per day.
Upper limb function | 15 minutes
  Disabilities of the Arm, Shoulder and Hand (DASH) - Scores 0 to 100. Higher the score worse the functionality of the upper limb.
Muscular Strength | 15 minutes
  Chatillôn® Portable Digital Dynamometer - Maximal force in Newton.
Range of motion | 15 minutes
  Carci goniometer - Maximal Angle
Posture | 10 minutes
  Postural evaluation - Postural alterations; Hyperlordosis; Hyperkyphosis; Shoulder protrusion; Scoliosis; Pelvic anteversion; Valgus genus; Anterior head.
Flexibility | 10 minutes
  Sit and reach test - Wells Bank - Maximum of the line.
Balance | 15 minutes
  MINIBESTest Equilibrium Assessment Systems Test - Each item is scored on a four-point ordinal scale, in which zero is the worst performance and three best performance.
Lymphedema | 15 minutes
  Arm volume in centimeters
Cardiorrespiratory fitness | 30 minutes
  Submaximal incremental exercise test (85% of maximum heart rate - HRmax) will be performed using a cycle ergometer (Lode Excalibur Sport, Groningen, the Netherlands).

CONTACTS AND LOCATIONS:
Overall Officials: Leonessa Boing, MSc, Principal Investigator — University of the State of Santa Catarina; Adriana CA Guimarães, PhD, Study Director — University of the State of Santa Catarina; Tatiana B Fretta, Principal Investigator — University of the State of Santa Catarina
Locations (1):
- Santa Catarina State University, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boing L, de Bem Fretta T, Stein F, Lyra VB, Moratelli JA, da Silveira J, Dos Santos Saraiva PS, Bergmann A, Lynch BM, de Azevedo Guimaraes AC. Can mat Pilates and belly dance be effective in improving body image, self-esteem, and sexual function in patients undergoing hormonal treatment for breast cancer? A randomized clinical trial. Arch Womens Ment Health. 2023 Apr;26(2):141-151. doi: 10.1007/s00737-023-01294-4. Epub 2023 Jan 30. PMID 36715766
- [Derived] Boing L, Fretta TB, Lynch BM, Dias M, Rosa LMD, Baptista F, Bergmann A, Fausto DY, Bocchi Martins JB, Guimaraes ACA. Mat Pilates and belly dance: Effects on patient-reported outcomes among breast cancer survivors receiving hormone therapy and adherence to exercise. Complement Ther Clin Pract. 2023 Feb;50:101683. doi: 10.1016/j.ctcp.2022.101683. Epub 2022 Nov 5. PMID 36403344
- [Derived] Boing L, do Bem Fretta T, de Carvalho Souza Vieira M, Pereira GS, Moratelli J, Sperandio FF, Bergmann A, Baptista F, Dias M, de Azevedo Guimaraes AC. Pilates and dance to patients with breast cancer undergoing treatment: study protocol for a randomized clinical trial - MoveMama study. Trials. 2020 Jan 7;21(1):35. doi: 10.1186/s13063-019-3874-6. PMID 31910872